CLINICAL TRIAL: NCT05374356
Title: High Spinal Anesthesia and the Incidence of Delirium After Cardiac Surgery: a Randomized-controlled Feasibility Trial
Brief Title: High Spinal Anesthesia and the Incidence of Delirium After Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HS23755 B2020:026
Record Dates: First submitted 2022-04-13; First posted 2022-05-16 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2023-06

CONDITIONS: Post-Operative Confusion
Keywords: Cardiac surgery; Delirium; Spinal anesthesia
MeSH Terms: conditions — Delirium | interventions — Morphine; Bupivacaine; Glucose

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to either general anesthesia (GA) or HSA + GA.
Who Masked: Outcomes Assessor
Masking Description: All patients will be assessed by the study investigator for presence/absence of delirium on postoperative days 1,2 & 3, as well as routine nursing assessment by the delirium assessment tool CAM-ICU, routinely done by nursing staff. Chart reviews will be conducted to confirm any additional incidence of delirium. The data collectors will not be aware whether the patient had a spinal anesthetic or not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High spinal anesthesia (Active Comparator): 1. Spinal group: will receive high spinal anesthesia with hyperbaric bupivacaine (0.3 to 0.6 mgs/kg) + preservative free morphine (3 mcg/kg).
  2. Standard intraoperative monitors will include ECG, pulse oximetry, end-tidal CO2 and anesthetic gas measurement, quantitative EEG monitoring (BIS monitor), arterial line, central venous pressure line and any other monitor as clinically indicated.
  3. Conduct of the general anesthetic will not be protocolized. It will be a pragmatic study. The attending anesthesiologist will attempt to have a BIS score of 20- 40 during the operation.
  Interventions: Drug: Intrathecal bupivacaine and morphine
- Control group (No Intervention): 1. Standard intraoperative monitors will include ECG, pulse oximetry, end-tidal CO2 and anesthetic gas measurement, quantitative EEG monitoring (BIS monitor), arterial line, central venous pressure line and any other monitor as clinically indicated.
  2. Conduct of the general anesthetic will not be protocolized. It will be a pragmatic study. The attending anesthesiologist will attempt to have a BIS score of 20- 40 during the operation.

INTERVENTIONS:
Drug: Intrathecal bupivacaine and morphine — Spinal group: will receive high spinal anesthesia with hyperbaric bupivacaine (0.3 to 0.6 mgs/kg) + preservative free morphine (3 mcg/kg).
  Other Names: Drug: bupivacaine 0.75% in dextrose (0.3 to 0.6 mls/kg); Drug: preservative free morphine 3 mcg/kg
  Arms: High spinal anesthesia

SUMMARY:
This is a feasibility study to determine if enough patients undergoing elective or urgent cardiac surgery, can be enrolled in a study where patients are randomized to receive high spinal anesthesia as an adjunct to general anesthesia for their cardiac surgery. The primary clinical outcome will be the incidence of post-operative delirium.

DETAILED DESCRIPTION:
Intervention

Patients will be randomized to either general anesthesia (GA) or HSA + GA.

1. Spinal group: will receive high spinal anesthesia with hyperbaric bupivacaine (0.3 to 0.6 mgs/kg) + preservative free morphine (3 mcg/kg).
2. Standard intraoperative monitors will include ECG, pulse oximetry, end-tidal CO2 and anesthetic gas measurement, quantitative EEG monitoring (BIS monitor), arterial line, central venous pressure line and any other monitor as clinically indicated.
3. Conduct of the general anesthetic will not be protocolized. It will be a pragmatic study. The attending anesthesiologist will attempt to have a BIS score of 20- 40 during the operation.
4. Intraoperative physiological data (mean blood pressure, end-tidal anesthetic gas concentrations, BIS score) will be recorded and downloaded to a laptop computer using the Trend Face Solo acquisition system for subsequent analysis.
5. The routine postoperative care map for the postoperative cardiac intensive care unit (ICCS) will be followed.
6. All patients will be assessed by the study investigator for presence/absence of delirium on postoperative days 1,2 & 3, as well as routine nursing assessment by the delirium assessment tool CAM-ICU, routinely done by nursing staff. Chart reviews will be conducted to confirm any additional incidence of delirium.
7. All patients will be contacted at one and three months after surgery and asked to complete a ten-minute survey (Postop QoR-15 questionnaire) assessing their quality of recovery.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 years old) patients
* Undergoing elective or urgent cardiac surgical procedures with cardiopulmonary bypass

Exclusion Criteria:

* Contraindications to spinal anesthesia such as active anticoagulation, clopidogrel within 7 days of surgery, ticagrelor within 3 days of surgery and all other contraindications to lumbar puncture
* Pre-existing psychiatric diagnoses such as schizophrenia or manic-depressive disorder
* Complex aortic surgery (> hemi-arch repair, descending thoracic surgery)
* Difficult airway requiring an awake intubation
* BMI > 50

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | One year
  Mean number of patients recruited per week) (n)
Protocol adherence measure - establishment of spinal anesthetic | Day of surgery
  In order to assess protocol adherence (%), in patients randomized to spinal anesthesia, an 80% success rate in establishing a spinal anesthetic will be considered as protocol adherence.
Protocol adherence measure - completion of delirium assessments | Day of surgery until five days post-operatively
  In order to assess protocol adherence (%), completion of 90% of scheduled delirium assessments will be considered protocol adherence.

SECONDARY OUTCOMES:
Early incidence of post-operative delirium | Day of surgery until five days post-operatively
  Duration of delirium (days) as assessed by the number of positive Confusion Assessment Method (CAM) as assessed by study investigator
Verification of early incidence of post-operative delirium | Day of surgery until five days post-operatively
  Duration of delirium (days) as assessed by the number of positive CAM Scores as assessed by nursing/physicians (by chart review).
Late incidence of post-operative delirium | Post-operative day 6 until post-operative day 14 or discharge from hospital whichever occurs first.
  Duration of delirium (days) as assessed by the number of positive CAM scores as assessed by study investigator from post-operative day 6 to post-operative day 14 or discharge from hospital
Verification of late incidence of post-operative delirium | Post-operative day 6 until post-operative day 14 or discharge from hospital, whichever occurs first.
  Duration of delirium (days) as assessed by the number of positive CAM scores as assessed by nursing/physicians (by chart review) from post-operative day 6 to discharge from hospital
Use of haloperidol post-operatively | Day of surgery until post-operative day 14 or discharge from hospital, whichever occurs first.
  Incidence (%) and total dose of haloperidol, in milligrams, for treatment of agitation as ordered by attending medical staff from day of surgery to discharge from hospital
Use of quetiapine post-operatively | Day of surgery until post-operative day 14 or discharge from hospital, whichever occurs first.
  Incidence (%) and total dose of quetiapine, in milligrams, for treatment of agitation as ordered by attending medical staff from day of surgery to discharge from hospital.
Use of risperidone post-operatively | Day of surgery until post-operative day 14 or discharge from hospital, whichever occurs first.
  Incidence (%) and total dose of risperidone, in milligrams, for treatment of agitation as ordered by attending medical staff from day of surgery to discharge from hospital.
Use of dexmedetomidine post-operatively | Day of surgery until post-operative day 5 or discharge from the intensive care unit whichever comes first..
  Incidence (%) of use of dexmedetomidine infusions, for treatment of agitation as ordered by attending medical staff from day of surgery to discharge from the intensive care unit.

OTHER OUTCOMES:
Incidence of intraoperative extubation | Day of surgery
  Incidence of extubation in the operating room (%)
Duration of ICU intubation | Day of surgery until post-operative day 14 or discharge from hospital, whichever occurs first.
  Duration of ICU intubation in hours for those patients brought intubated to the ICU
Post-operative pain scores at rest | Post-operative day 1 until post-operative day 3
  VAS pain scores (visual analog score) (0 is no pain, 10 is the worst pain possible) at rest for 3 days post-operatively.
Post-operative pain scores with deep breathing | Post-operative day 1 until post-operative day 3
  VAS pain scores (0 is no pain, 10 is the worst pain possible) with deep breathing for 3 days post-operatively.
Post-operative hydromorphone administered | Day of surgery until post-operative day 3
  Total hydromorphone use including intravenous and oral administration will be recorded for the first 48 hours postoperatively. Hydromorphone totals will be converted to morphine equivalents using MD Calcs algorithm (https://www.mdcalc.com/morphine-milligram-equivalents-mme-calculator).
Post-operative fentanyl administered | Day of surgery until post-operative day 3
  Total fentanyl use including intravenous and oral administration will be recorded for the first 48 hours postoperatively. Fentanyl totals will be converted to morphine equivalents using MD Calcs algorithm (https://www.mdcalc.com/morphine-milligram-equivalents-mme-calculator).
Post-operative codeine administered | Day of surgery until post-operative day 3
  Total codeine use including intravenous and oral administration will be recorded for the first 48 hours postoperatively. Codeine totals will be converted to morphine equivalents using MD Calcs algorithm (https://www.mdcalc.com/morphine-milligram-equivalents-mme-calculator).
Post-operative morphine administered | Day of surgery until post-operative day 3
  Total morphine use, in milligrams, including intravenous and oral administration will be recorded for the first 48 hours postoperatively.
Intraoperative hypotension | Day of surgery
  Length of time (mins) mean arterial blood pressure is less than 55 mmHg
Intraoperative end-tidal gas concentration | Day of surgery
  Mean intraoperative end-tidal gas concentration (%)
Intraoperative depth of anesthesia | Day of surgery
  Mean intraoperative bispectral index (BIS). The BIS scale range is from 0 to 100, with 0 representing no measurable electrical brain activity and 100 the electrical activity of an awake, conscious individual. Currently BIS scores are attempted to be kept between 20 and 40 during surgery to ensure adequate depth of anesthesia.
Intraoperative sufentanil administered | Day of surgery
  Total dose of intraoperative sufentanil in micrograms. Sufentanil dosage will be converted to morphine equivalents using the MD Calcs algorithm (https://www.mdcalc.com/morphine-milligram-equivalents-mme-calculator)
Intraoperative hydromorphone administered | Day of surgery
  Total dose of intraoperative hydromorphone in milligrams. Hydromorphone doses will be converted to morphine equivalents using the MD Calcs algorithm (https://www.mdcalc.com/morphine-milligram-equivalents-mme-calculator)
Intraoperative midazolam administered | Day of surgery
  Total dose of intraoperative midazolam in milligrams.
Intraoperative ketamine administered | Day of surgery
  Total dose of intraoperative ketamine in milligrams
Intraoperative glucose level | Day of surgery
  Highest intraoperative glucose level in millimoles per litre.
Intraoperative insulin administered | Day of surgery
  Total intraoperative insulin administered in units of insulin.
Total RBC utilization | Day of surgery until post-operative day 3
  Total RBC administered (units) both intraoperatively, and postoperatively until post-operative day 3..
Total platelet utilization | Day of surgery until post-operative day 3
  Total units of platelets administered (adult doses of platelets ) both intraoperatively, and postoperatively until post-operative day 3
Return to OR for bleeding | Day of surgery until post-operative day 3
  Incidence of a return to the operating room for bleeding (%)
Vasopressor (norepinephrine or phenylephrine or vasopressin) use at 12 hours | First 12 hours postoperatively
  Incidence of use of either norepinephrine, phenylephrine or vasopressin at 12 hours postoperatively (%)
Vasopressor (norepinephrine, phenylephrine or vasopressin) use at 24 hours | 12 to 24 hours postoperatively
  Incidence of use of norepinephrine, phenylephrine or vasopressin administered at 24 hours postoperatively (%)
Vasopressor (norepinephrine, phenylephrine or vasopressin) use at >24 hours | Post-operative day 2 to post-operative day 7
  Incidence of norepinephrine, phenylephrine or vasopressin use longer than 24 hours postoperatively (%)
Incidence of re-intubation | Day of surgery until 14 days post-operatively or discharge from hospital, whichever occurs first.
  Incidence of re-intubation postoperatively (%) from day of surgery to discharge from hospital
ICU re-admission | Post-operative day 2 until post-operative day 14 or discharge from hospital, whichever occurs first.
  Incidence of re-admission to ICU for any reason from post-operative day 2 to post-operative day 14 or discharge from hospital (%)
Hospital length of stay | Time (days) in hospital from post-operative 1 to 30 (or through discharge from hospital)
  Postoperative hospital length of stay in days
ICU length of stay | Time (days) in ICU from post-operative day 1 to 5 (or through discharge from hospital)
  Postoperative ICU length of stay in days
Major medical complications | Day of surgery until post-operative day 14 or discharge from hospital, whichever occurs first.
  Incidence of major medical complications (%) defined as one or more of: a. Atrial fibrillation b. Pneumonia c. Acute kidney injury (defined as a doubling of pre-operative creatinine) d. Need for dialysis e. Wound infection f. Stroke g. Other
Post-operative quality of recovery - one month | 30 days post surgery
  Postoperative quality of life score (Postop QoR-15) will be used to assess quality of recovery at one month postoperatively. The Post QoR-15 scale ranges from 0 to 150, with 0 representing the poorest quality of recovery and 150 the best quality of recovery.
Post-operative quality of recovery - three months | 90 days post surgery
  Postoperative quality of life score (Postop QoR-15) will be used to assess quality of recovery at three month postoperatively. The Post QoR-15 scale ranges from 0 to 150, with 0 representing the poorest quality of recovery and 150 the best quality of recovery.
Post-operative creatinine level | Day of surgery until 14 days post-operatively or hospital discharge, whichever occurs first.
  Highest post-operative creatinine (umol/l) level recorded during hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Doug Maguire, MD, Study Director — University of Manitoba
Locations (1):
- St. Boniface Hospital, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No